CLINICAL TRIAL: NCT00837928
Title: Phase I Study of Bendamustine and Fractionated Stereotactic Radiotherapy of Patients With 1- 4 Brain Metastases From Solid Malignancies
Brief Title: Bendamustine and Radiation Therapy in Treating Patients With Brain Metastases Caused by Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Grecula (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor-Investigator, John Grecula, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08142; NCI-2011-03179 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Bendamustine Hydrochloride; Surgical Procedures, Operative; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine and Fractionated stereotactic radiotherapy (Experimental): Bendamustine 40 mg/m2 and will be administered IV on days 1,2,and 3 prior to surgery on each day of SRT (Sterotactic radiation therapy). Laboratory biomarker analysis will be obtained on day 1 or 2 only from patients undergoing surgery on day 3 (i.e. Pharmacokinetic samples will not be collected from patients who begin SRT on day 1). Surgical Resection of Brain Metastases Day 3 (immediately after Bendamustine) Stereotactic fractionated radiation therapy starting at least 4 weeks after surgery (Day 1 if no surgery ); 30 Gy in 5 daily fractions(Mon-Fri). Concurrent Bendamustine is administered on Days of Stereotactic Radiotherapy (Arm 1: 40 mg/m2/ Day; Arm 2: 50 mg/m2/day).
  Interventions: Drug: bendamustine; Other: laboratory biomarker analysis; Procedure: Surgical Resection of Brain Metastases; Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Drug: bendamustine — 40 mg/m2 will be administered IV on days 1,2,and 3 prior to surgery.on each day of SRT.
  Other Names: Ribomustin; Treanda
Other: laboratory biomarker analysis — samples will be obtained on day 1 or 2 only from patients undergoing surgery on day 3 (i.e. PK samples will not be collected from patients who begin SRT on day 1).
  Other Names: Laboratory Procedure
Procedure: Surgical Resection of Brain Metastases — Surgical Resection of Brain Metastases Day 3 (immediately after Bendamustine)
  Other Names: surgery
Radiation: Stereotactic body radiation therapy — Starting at least 4 weeks after surgery (Day 1 if no surgery ); 30 Gy in 5 daily fractions(Mon-Fri)
  Other Names: SRT; Stereotactic Fractionated Radiation Therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bendamustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of bendamustine when given together with radiation therapy in treating patients with brain metastases caused by solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the recommended phase II dose of bendamustine hydrochloride when administered in combination with stereotactic radiotherapy for the treatment of patients with 1-4 brain metastases from solid malignancies.

Secondary

* Determine bendamustine hydrochloride pharmacokinetics and correlate this to bendamustine hydrochloride levels in brain metastases, brain margin, arachnoid, cerebral spinal fluid, and plasma acquired at the time of surgery.
* Assessment of local control of brain metastases.

OUTLINE: This is a dose-escalation study of bendamustine hydrochloride.

Patients with no potentially resectable lesion(s) receive bendamustine hydrochloride IV over 30 minutes and stereotactic radiotherapy once daily for 5 days.

Patients with potentially resectable lesion(s) receive bendamustine hydrochloride IV over 30 minutes on days 1-3 and undergo surgery on day 3. At least 4 weeks after surgery, these patients receive adjuvant bendamustine hydrochloride and stereotactic fractionated radiotherapy as above (in patients with no potentially resectable lesion[s])

Blood samples are collected periodically for pharmacokinetic studies. Cerebrospinal fluid, arachnoid, tumor margin, and tumor samples are also collected during surgery for correlative studies.

After completion of study treatment, patients are followed every 3 months for 21 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer with 1 to 4 brain metastases imaged by MRI/CT scans not involving thalamus, basal ganglia or brain stem.
* No cancer originating in central nervous system
* Candidate for clinically indicated surgery to resect brain lesions.
* Karnofsky score of at least 60
* At least 18 years of age
* Life expectancy of more than two months

Exclusion Criteria:

* Evidence of leptomeningeal metastases.
* Need immediate treatment to prevent neurological deterioration.
* Prior brain radiotherapy or surgery for current brain metastases.
* Radiosensitive primary tumors such as small cell lung cancer, germ cell tumors, lymphoma, leukemia or multiple myeloma.
* Absolute neutrophil count (ANC)<1500/mm3 or platelets <50,000/mms.
* Brain metastasis diameter greater than 5 cm.
* Not pregnant or nursing
* More than 3 weeks since prior chemotherapy.
* No evidence of ischemia on EKG and/or reduced cardiac ejection fraction (i.e., < 50%) on ECHO.
* No known sensitivity or allergy to bendamustine hydrochloride or mannitol
* No more than 3 prior cytotoxic chemotherapy regimens
* No unresolved persistent toxicities for 4 weeks from prior chemotherapy or 6 weeks for nitrosoureas.
* Calculated creatinine clearance <40 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02-19 (Actual); Primary Completion 2015-01-08 (Actual); Study Completion 2015-01-08 (Actual)

PRIMARY OUTCOMES:
Determine recommended dose of Bendamustine when used in combination with Stereotactic Radiotherapy (STR) for treatment of patients with 1-4 brain metastases. | up to 4 years

SECONDARY OUTCOMES:
Pharmacokinetics of bendamustine | up to 4 years
Levels of bendamustine hydrochloride in the brain metastases, brain margin, arachnoid, cerebral spinal fluid, and plasma | up to 4 years
Local control of brain metastases | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: John C. Grecula, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu